CLINICAL TRIAL: NCT03753451
Title: Influence of Periodontal Disease Treatment on Serum Levels of Sirtuin 1 and Mannose-binding Lectin in Individuals With Coronary Artery Disease
Brief Title: Influence of Periodontal Disease Treatment on Serum Levels of Sirtuin 1 and Mannose-binding Lectin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InCor Heart Institute (Other)
Responsible Party: Principal Investigator, ANTONIO DE PADUA MANSUR, Principal Investigator, InCor Heart Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDC 4329/15/156
Record Dates: First submitted 2018-11-06; First posted 2018-11-27 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Periodontal Diseases
Keywords: periodontal diseases; atherosclerosis; mannose binding protein; sirtuins; inflammation
MeSH Terms: conditions — Periodontal Diseases; Atherosclerosis; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (No Intervention): 20 patients without periodontal disease and coronary artery disease
- Group 2 (No Intervention): 20 patients without periodontal disease and with coronary artery disease
- Group 3 (Active Comparator): 20 patients with periodontal disease and with coronary artery disease received treatment of periodontal disease
  Interventions: Procedure: treatment of periodontal disease
- Group 4 (Active Comparator): 20 patients with periodontal disease and without coronary artery disease received treatment of periodontal disease
  Interventions: Procedure: treatment of periodontal disease

INTERVENTIONS:
Procedure: treatment of periodontal disease — Patients with periodontal disease received treatment of periodontal disease through ultrasound or manual scaling of dental calculations. In addition to receiving instructions to improve oral health, such as the correct use of dental floss, adequate time and the correct way to brush.
  Arms: Group 3; Group 4

SUMMARY:
The premise of the relationship between the atherosclerotic process of coronary artery disease and periodontal disease is the immunoinflammatory process, which causes a significant increase in serum concentration of mannose-binding lectin. This protein is part of the innate immunity and has the ability to bind to the mannose residues common to various pathogens. Animal studies also showed that increased serum concentration of sirtuin-1 was associated with reduced inflammation. Evidence indicates that sirtuin-1 plays an important role in vascular protection and is associated with aging. OBJECTIVES: This study examined the influence of non-surgical treatment of periodontal disease on the serum concentration of mannose-binding lectin and sirtuin-1 in patients with periodontal disease and coronary artery disease. METHODS: Seventy-eight patients, 38 women and 40 men, mean age 58 ± 8 years old, were divided into 4 groups: 20 healthy subjects (group 1), 18 patients with coronary artery disease and without periodontal disease (group 2), 20 patients with periodontal disease and without coronary artery disease (group 3) and 20 patients with coronary artery disease and periodontal disease (group 4). Peripheral blood samples were collected at the beginning and at the end of the treatment of periodontal disease.

DETAILED DESCRIPTION:
Inclusion criteria for PD were: presence of at least 15 teeth and clinical diagnosis of PD. Excluding third molars. This diagnosis was confirmed by the presence of at least 6 teeth with at least one noncontiguous interproximal site with Probing Pocket Depth (PPD) and Clinical Attachment Loss (CAL) ≥ 5 mm, as well as 30% of Sites with PPD and CAL ≥ 4mm and bleeding on Probing (BOP). Periodontal disease currently classified as Stage III Degree B. Periodontal healthy was defined as individuals who presented a periodontium without loss of insertion, with PPD ≤3 mm, BOP in less than 10% of the sites and without radiographic bone loss.

Non-surgical periodontal treatment was performed, including oral hygiene education, scaling, smoothing and coronal-radicular polishing (RAR). Six sites were evaluated in each tooth (mesiobuccal, buccal, distobuccal, distolingual/palatal, lingual/palatal and mesiolingual/palatal surfaces). Scaling and root planing were performed using mechanical devices - ultrasound and manual instruments. The treatment was with local anesthesia, 3% lidocaine with vasoconstrictor, for PPD ≥ 5 mm. The objective of each session was to achieve a smooth surface, devoid of biofilm and calculus.

The following parameters are evaluated during clinical examination: Probing Pocket Depth (PPD), distance of the enamel-cementum line at the gingival margin, clinical Attachment Loss (CAL), plaque index (IP) and bleeding on probing (BOP), PPD and CAL measurements are rounded to the nearest millimeter using a North Carolina periodontal probe (Chicago, USA).

ELIGIBILITY:
Inclusion Criteria:

* Presence of installed periodontal disease.
* More than 15 teeth in the mouth

Exclusion Criteria:

* uncontrolled diabetic,
* dialytic,
* smokers,
* patients with HIV and Hepatitis B and C.
* Pregnant subjects,
* edentulous patients,
* orthodontic brachytherapy were excluded from the study,
* patients using specific drugs known to affect periodontal tissues,
* patients who have undergone previous periodontal treatment (minimum of 6 months), * patients taking anti-inflammatory drugs and corticosteroids.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
After improving the periodontal clinical aspects, we observed whether there was an impact on serum levels of mannose-binding lectin (MBL) protein. | The periodontal treatment was performed and at the end of three-month period blood sample was collected.
  Non-surgical periodontal treatment was performed to treat the periodontal disease and it included oral hygiene education, scaling, smoothing and polishing of the root and dental crown (RAR). Blood sample was collected at baseline and at the end of study.
After improving the periodontal clinical aspects, we observed whether there was an impact on serum levels of sirtuin-1 (SIRT1) protein. | The periodontal treatment was performed and at the end of three-month period blood sample was collected.
  Non-surgical periodontal treatment was performed to treat the periodontal disease and it included oral hygiene education, scaling, smoothing and polishing of the root and dental crown (RAR). Blood sample was collected at baseline and at the end of study.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio P Mansur, 1, Principal Investigator — Universidade de São Paulo, São Paulo, SP, BR
Locations (2):
- Brazil (2):
  - INCOR- Heart Institute, São Paulo, São Paulo
  - INCOR - Heart Institute, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mansur AP, Roggerio A, Goes MFS, Avakian SD, Leal DP, Maranhao RC, Strunz CMC. Serum concentrations and gene expression of sirtuin 1 in healthy and slightly overweight subjects after caloric restriction or resveratrol supplementation: A randomized trial. Int J Cardiol. 2017 Jan 15;227:788-794. doi: 10.1016/j.ijcard.2016.10.058. Epub 2016 Oct 27. PMID 28029409
- [Result] Liukkonen A, He Q, Gursoy UK, Pussinen PJ, Grondahl-Yli-Hannuksela K, Liukkonen J, Sorsa T, Suominen AL, Huumonen S, Kononen E. Mannose-binding lectin gene polymorphism in relation to periodontal infection. J Periodontal Res. 2017 Jun;52(3):540-545. doi: 10.1111/jre.12420. Epub 2016 Sep 14. PMID 27624657
- [Result] Tsutsumi A, Kobayashi T, Ito S, Goto D, Matsumoto I, Yoshie H, Sumida T. Mannose binding lectin gene polymorphism and the severity of chronic periodontitis. Nihon Rinsho Meneki Gakkai Kaishi. 2009 Feb;32(1):48-52. doi: 10.2177/jsci.32.48. PMID 19252378
- [Result] Louropoulou A, van der Velden U, Schoenmaker T, Catsburg A, Savelkoul PH, Loos BG. Mannose-binding lectin gene polymorphisms in relation to periodontitis. J Clin Periodontol. 2008 Nov;35(11):923-30. doi: 10.1111/j.1600-051X.2008.01311.x. Epub 2008 Sep 20. PMID 18823346
- [Result] Mattagajasingh I, Kim CS, Naqvi A, Yamamori T, Hoffman TA, Jung SB, DeRicco J, Kasuno K, Irani K. SIRT1 promotes endothelium-dependent vascular relaxation by activating endothelial nitric oxide synthase. Proc Natl Acad Sci U S A. 2007 Sep 11;104(37):14855-60. doi: 10.1073/pnas.0704329104. Epub 2007 Sep 4. PMID 17785417

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/51/NCT03753451/Prot_SAP_000.pdf
  • Informed Consent Form (2016-10-06): https://cdn.clinicaltrials.gov/large-docs/51/NCT03753451/ICF_001.pdf